CLINICAL TRIAL: NCT01165112
Title: A Phase I/II Trial of Bendamustine/Treanda®, Rituximab, Etoposide, and Carboplatin for Patients With Relapsed or Refractory Lymphoid Malignancies and Select Untreated Lymphomas (TREC)
Brief Title: Bendamustine Hydrochloride, Rituximab, Etoposide, and Carboplatin in Treating Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma or Hodgkin Lymphoma
Acronym: TREC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Gopal, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSOC 2502; NCI-2010-00907 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PSOC 2502 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2010-06-21; First posted 2010-07-19 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease | interventions — Bendamustine Hydrochloride; Carboplatin; Rituximab; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy and monoclonal antibody therapy) (Experimental): Patients receive bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2, etoposide IV over 60 minutes on days 1-3, and carboplatin IV over 60 minutes on day 1. Patients with CD20+ T-cell lymphoma disease also receive rituximab IV on day 2 or 3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bendamustine Hydrochloride; Drug: Carboplatin; Biological: Rituximab; Drug: Etoposide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Ribomustin; SyB L-0501; Treanda
Drug: Carboplatin — Given IV
Biological: Rituximab — Given IV
  Other Names: MOAB IDEC-C2B8
Drug: Etoposide — Given IV
  Other Names: Lastet
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of bendamustine hydrochloride when given together with carboplatin, etoposide, and rituximab in treating patients with diffuse large B cell lymphoma or Hodgkin lymphoma that has come back after a period of improvement or has not responded to previous treatment. Drugs used in chemotherapy, such as bendamustine hydrochloride, etoposide, and carboplatin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, may block cancer growth by targeting certain cells. Giving bendamustine hydrochloride together with carboplatin, etoposide, and rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximally tolerated dose of bendamustine (bendamustine hydrochloride) that can be combined with rituximab, carboplatin, and etoposide chemotherapy in patients with relapsed or refractory lymphoid malignancies.

II. To determine the safety and toxicity of the above regimen.

SECONDARY OBJECTIVES:

I. To gain a preliminary assessment of the efficacy of the above regimen.

II. To determine the ability to proceed to peripheral blood stem cell collection following the above regimen (the impact of above regimen on stem cell reserve).

III. To investigate whether findings from laboratory, radiographic or pathologic studies have any prognostic impact on the response to treatment.

OUTLINE: This is a phase I, dose-escalation study of bendamustine hydrochloride followed by a phase II study.

Patients receive bendamustine hydrochloride intravenously (IV) over 30-60 minutes on days 1 and 2, etoposide IV over 60 minutes on days 1-3, and carboplatin IV over 60 minutes on day 1. Patients with cluster of differentiation (CD)20+ T-cell lymphoma disease also receive rituximab IV on day 2 or 3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have relapsed or primary refractory lymphomas: diffuse large B cell lymphoma (DLBCL) or Hodgkin's lymphoma (HL); patients with other lymphoid malignancies such as T- cell, or lymphomas that are not curable with anthracycline based therapy (e.g. mantle cell lymphoma [MCL], follicular lymphoma [FL], marginal zone lymphoma [MZL], lymphoplasmacytic lymphoma [LPL]) are eligible with protocol Chair review and approval; Note: as of 11/1/12 only patients with typical DLBCL and HL are eligible for enrollment; unusual pathology for DLBCL and HL will require Study Chair approval; the goal is to have 20 patients with DLBCL and 20 patients with HL enrolled
* World Health Organization (WHO) classification of patient's malignancies must be provided
* Patients must have measurable disease defined as lesions that can be accurately measured in two dimensions by computed tomography (CT), magnetic resonance imaging (MRI), medical photograph (skin or oral lesion), plain x-ray, or other conventional technique and a greatest transverse diameter of 1 cm or greater; or palpable lesions with both diameters >= 2 cm; Note: CT scans remain the standard for evaluation of nodal disease
* Patients must have a CT of chest, abdomen, and pelvis within 28 days of enrollment; patients with evidence of lymphadenopathy in the neck must have a CT of neck
* Patients should not have evidence of active central nervous system lymphoma
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,500/mm^3 (without transfusion or growth factor support); exception: patients with cytopenias due to disease, that do not meet these criteria, will be considered eligible with review and approval by the principal investigator (PI) or Co-PI prior to study entry
* Platelets >= 100,000/mm^3 (without transfusion or growth factor support); exception: patients with cytopenias due to disease, that do not meet these criteria, will be considered eligible with review and approval by the PI or Co-PI prior to study entry
* Serum creatinine < 1.5 mg/dl or creatinine clearance greater than 50/ml per minute
* Total bilirubin < 1.5 times upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal
* Patients must have a serum lactate dehydrogenase (LDH) performed within 14 days prior to registration
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines
* Patients must be anticipated to complete at least 2 cycles of chemotherapy

Exclusion Criteria:

* Patients known positive for human immunodeficiency virus (HIV), or infectious hepatitis type B or C
* Pregnant or nursing women; men or women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients with other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, breast or cervical cancer in situ, or other cancer from which the patient has been disease-free for 5 years or greater, unless approved by the protocol Chair
* Patients who are refractory (i.e. not responded or progressed within 6 months) to a carboplatin, cisplatin, bendamustine, or etoposide-based regimen
* Patients who have other medical conditions that would contraindicate treatment with aggressive chemotherapy (including active infection, uncontrolled hypertension, congestive heart failure, unstable angina pectoris, or myocardial infarction within the past 6 months, uncontrolled arrhythmia); if the patient's cardiac history is questionable, a measurement of left ventricular ejection fraction should be obtained within 42 days prior to registration; patients with left ventricular ejection fraction < 50% are not eligible
* Autologous or allogeneic transplantation within 12 months or radioimmunotherapy within 6 months of registration; prior failed (< 5 x 10^6 CD34/kg) peripheral blood stem cell (PBSC) collection
* Patients who had pelvic radiation within 12 months or received more than 2 prior therapies with myelotoxic regimens; single agent monoclonal antibody treatment is not considered as one therapy; radiation treatment following chemotherapy is not considered as one separated therapy; consolidative therapy will be considered one regimen e.g. salvage therapy followed by conditioning regimen and transplant
* Previous chemotherapy/immunotherapy within 3 weeks before study entry
* Concurrent use of other anti-cancer agents or experimental treatments
* Known hypersensitivity to bendamustine, mannitol, etoposide, carboplatin, or rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Budde LE, Wu D, Martin DB, Philip M, Shustov AR, Smith SD, Gooley TA, Chen TL, Libby EN, Chen EY, Kojouri K, Langerak A, Roden JE, Press OW, Gopal AK. Bendamustine with rituximab, etoposide and carboplatin (T(R)EC) in relapsed or refractory aggressive lymphoma: a prospective multicentre phase 1/2 clinical trial. Br J Haematol. 2018 Nov;183(4):601-607. doi: 10.1111/bjh.15585. Epub 2018 Sep 14. PMID 30596402

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy and Monoclonal Antibody Therapy)
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy and Monoclonal Antibody Therapy)
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 56 [23 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 43
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose of Bendamustine Hydrochloride That Can be Combined With Rituximab, Carboplatin, and Etoposide Chemotherapy in Patients With Relapsed or Refractory Lymphoid Malignancies
Description: Defined as dose at which approximately =< 25% of patients experience a DLT. Following completed observation of final patient, two-parameter logistic model fit to data, generating dose-response curve based on observed toxicity rate at dose levels visited. Based on this fitted model, MTD is estimated to be dose that is associated with toxicity rate of 25%. If estimate of slope parameter for fitted curve is not positive and finite, geometric mean of dose level used for last cohort and dose level that would have been assigned to next cohort is taken as MTD.
Time Frame: Up to 5 weeks after the last course
Measure: Number; unit: mg/m2 x 2
Arm/Group | Treatment (Chemotherapy and Monoclonal Antibody Therapy)
Number analyzed (Participants) | 48
mg/m2 x 2 | 120

2. Primary Outcome: Safety and Toxicity of This Regimen
Description: Count of participants experiencing a dose limiting toxicity. The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0 will be used to classify and grade toxicities.
Time Frame: Up to 5 weeks after the last course
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Monoclonal Antibody Therapy)
Number analyzed (Participants) | 48
Participants | 0

3. Secondary Outcome: Preliminary Assessment of the Efficacy of This Regimen
Description: Response will be defined by standard NCI criteria (Cheson et al) for lymphoid malignancies.
Time Frame: Up to 5 weeks after the last course
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Monoclonal Antibody Therapy)
Number analyzed (Participants) | 47
Participants | 33

4. Secondary Outcome: Ability to Proceed to Peripheral Blood Stem Cell (PBSC) Collection Following Treatment (Impact of This Regimen on Stem Cell Reserve)
Time Frame: Up to 5 weeks after the last course
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Monoclonal Antibody Therapy)
Number analyzed (Participants) | 32
Participants | 30

ADVERSE EVENTS:
Arm/Group | Treatment (Chemotherapy and Monoclonal Antibody Therapy)
Serious Adverse Events (participants affected / at risk) | 14/48
Other Adverse Events (participants affected / at risk) | 46/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy and Monoclonal Antibody Therapy) (N=48)
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Catheter related infection (Infections and infestations) | 1
Obstruction gastric (Gastrointestinal disorders) | 2
Allergic reaction (Immune system disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Fever (General disorders) | 2
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Aseptic Meningitis (Infections and infestations) | 1
Vascular access complication (Vascular disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy and Monoclonal Antibody Therapy) (N=48)
Anemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 30
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 4
Infection (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes